CLINICAL TRIAL: NCT05144750
Title: Fruit and Vegetable Prescription in the Community Health Center Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wholesome Wave (Other)
Collaborators: One Community Health (Unknown); Yale-Griffin Prevention Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000030975
Record Dates: First submitted 2021-11-03; First posted 2021-12-03 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Poverty
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruit and Vegetable Prescription Program Cohort (Experimental): All participants received the program intervention.
  Interventions: Behavioral: Fruit and Vegetable Prescription

INTERVENTIONS:
Behavioral: Fruit and Vegetable Prescription — The intervention adds a $50 monthly fruit and vegetable voucher, and text reminder and educational text messages (recipes/tips) to the Standard of Care for patients.
  Standard Care for Patients at OCH: Patients will be able to regularly meet with their healthcare team.
  Fruit and Vegetable Incentive: During the 8-month intervention period, registered program participants can receive $50 monthly through the reloadable Walmart gift card, which can only be used to purchase fresh fruits and vegetables. The total incentive will be $400 for the eight-month program.
  Text Communication: Wholesome Wave will share text reminders to shop and utilize incentives. Wholesome Wave will also share text messages that are consistent with the messages that the OCH dietitians are offering in their standard care, including recipes and tips.
  Other Names: Fruit and Vegetable Incentive

SUMMARY:
The proposed study examines the implementation and efficacy of a fruit and vegetable incentive program in a population of adults with diabetes at a community health center (CHC) in California. Additionally, we seek to understand the impact of this program on the participants with particular attention to their experience and point of view. To better understand the program and its impact, a mixed methods approach will be used.

DETAILED DESCRIPTION:
The proposed research will utilize a mixed methods approach with both qualitative and quantitative methods to assess the process and impact of a fruit and vegetable incentive program administered in a community clinic that serves a population that is low-income in Sacramento, California.

Sacramento County has a population of 1.5 million people and 500,000 people living in the city of Sacramento proper. The poverty rate of the county over all is 12.6% and the city is 16.6%. The most recent estimate of county level food insecurity is 12%, which is consistent with the national average; however, the estimated rate during the COVID 19 pandemic is 16.5%. Sacramento also serves as an ideal region for intervention because there is a strong community partner with the CHC, One Community Health (OCH) and there are regionally accessible Walmart stores at which the fruit and vegetable incentives (i.e., Walmart gift cards) can be used. Participants in the study will receive up to $400 in fruit and vegetable vouchers over 8 months, $50 in voucher given per household each month (paused if no voucher redemption within prior 2 months).

The intervention adds a $50 monthly fruit and vegetable voucher, and text reminder and educational text messages (recipes/tips) to the Standard of Care for patients.

Standard Care for Patients at OCH: Patients/participants will be able to regularly meet with their healthcare team which includes but is not limited to a primary care physician, nursing staff, dietitians and other providers as needed. All care is based on evidence-based best clinical practices and the patient's voluntary involvement with their providers.

Fruit and Vegetable Incentive: During the 8-month intervention period, registered program participants can receive $50 monthly through the reloadable Walmart gift card, which can only be used to purchase fresh fruits and vegetables. The total incentive will be $400 for the eight-month program. Each month, program participants will be able to receive their monthly $50 incentive, providing their balance at the time of the reload does not exceed $100, due to two months of inactivity. Monthly reload plan will be made based on available balance during the first week of each month, with the reload planned for the 15th of each month.

Text Communication: Participants will share a text-enabled phone number with Wholesome Wave for Wholesome Wave to send text reminders to shop and utilize incentives, likely 2 times per month. Wholesome Wave will also share text messages that are consistent with the messages that the OCH dietitians are offering in their standard care, including recipes and tips.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Low Income
* Patient of OCH

Exclusion Criteria:

* Under 18
* Does not speak Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index from Baseline to End of Program | All clinical measurements were collected at month 1 (baseline) and 8 (completion)
  Body mass index was calculated from height in meters and weight in kilograms: Height and Weight will be collected at months 1, 4 and 8 and at any additional clinic visits when appropriate.
  Weight and height will be combined to report BMI in kg/m^2
Change in HbA1c from Baseline to End of Program | All clinical measurements were collected at month 1 (baseline) to 8 (completion)
  Glycated hemoglobin A1c (HbA1c) was used to measure the average plasma glucose concentration. HbA1c will be measured using a finger-prick test. HbA1c will be reported as HbA1c% and Blood Glucose (mmol/L). Change in HbA1C will be calculated as end of program HbA1c% - baseline HbA1c%.
Glycemic Control | All clinical measurements were collected at month 1 (baseline) and 8 (completion)
  Glycemic control: Glycated hemoglobin A1c (HbA1c) will be used to measure the average plasma glucose concentration. HbA1c will be measured using a finger-prick test. HbA1c will be reported as HbA1c% and Blood Glucose (mmol/L). Glycemic control will be determined inline with American Diabetes Association guidelines. According to the ADA HbA1C values lower than 5.7% represents a normal range, between 5.7% and 6.5% is prediabetes and greater than 6.5% is diabetes.
Change in Blood Lipids HDL Ratio from Baseline to end of Program | All clinical measurements were collected at month 1 (baseline) and 8 (completion)
  Blood lipids: Values of total cholesterol (Tchol), triglycerides (TG), and high-density lipoprotein (HDL) will be obtained by clinical staff at OCH and run through their typical lab procedures that are part of standard of care, the values will be shared with researchers for months 1 and 8. HDL:Tchol ratio will also be computed. Change in HDL ration will be calculated as End of Program HDL ratio- beginning of the program HDL ratio.
Change in Blood Lipids LDL Ratio from Baseline to end of Program | All clinical measurements were collected at month 1 (baseline) and 8 (completion)
  Blood lipids: Values of total cholesterol (Tchol), triglycerides (TG), and high-density lipoprotein (HDL) will be obtained by clinical staff at OCH and run through their typical lab procedures that are part of standard of care, the values will be shared with researchers for months 1 and 8. Serum low-density lipoprotein (LDL) will be calculated using the following formula LDL = Tchol - (TG/5 + HDL). Change in LDL ratio will be calculated as End of Program LDL ratio- beginning of the program LDL ratio.
Change in Blood Pressure from Baseline to end of Program | All clinical measurements were collected at month 1 (baseline) and 8 (completion)
  Blood pressure: Blood pressure will be collected at by clinical staff at OCH at months 1 and 8 and at other clinical appointments as is medically appropriate, using an automatic blood pressure measurement device. Blood pressure will be measures as Systolic mm Hg/ diastolic mm Hg. Following the standards delineated by the CDC, systolic: less than 120 mm Hg diastolic: less than 80 mm Hg; systolic: 120-139 mm Hg diastolic: 80-89 mm Hg; and systolic: 140 mm Hg or higher diastolic: 90 mm Hg or higher. Change in blood pressure will be calculated change in (8 months systolic-1 month systolic) systolic over the change in diastolic (8 months diastolic-1 month diastolic).
Change in Food Security | Month 1(baseline) and 8 (completion)
  Food security will be measured using the USDA Household Food Security Measure. The score will be calculated following the USDA HFSM guide and change in food security will be reported as end of program score - beginning of program score.

SECONDARY OUTCOMES:
Fruit and Vegetable Consumption | Month 1(baseline) and 8 (completion)
  Fruit and vegetable consumption data will be measured using a short form fruit and vegetable food frequency questionnaire. The food frequency questionnaire will be scored and change in consumption will be calculated as end of program score - start of program score.
Self Reported Improved Health | Month 1(baseline) and 8 (completion)
  Self-reported improved health will be measured using the RAND single-item measure. Change in score will be calculated as change in mean.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Duffany, Principal Investigator — Yale University
Locations (1):
- One Community Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No